CLINICAL TRIAL: NCT02181387
Title: Does Acetaminophen Reduce Neuraxial Analgesic Requirement During Labor
Brief Title: Acetaminophen Use in Labor - Does Use of Acetaminophen Reduce Neuraxial Analgesic Drug Requirement During Labor?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: funding and compounding issues
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00023934
Record Dates: First submitted 2014-03-27; First posted 2014-07-03 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: labor pain; acetaminophen
MeSH Terms: conditions — Pain; Labor Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- acetaminophen (Active Comparator): 1000 mg every 6 hours during labor up to maximum 3 doses
  Interventions: Drug: Acetaminophen
- placebo (Placebo Comparator): placebo capsule identical to the acetaminophen capsule will be administered every 6 hours to a maximum of 4 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — administered every 6 hours by mouth up to 4 doses
  Other Names: tylenol
  Arms: acetaminophen
Drug: Placebo
  Arms: placebo

SUMMARY:
The hypothesis is if administration of acetaminophen during labor will reduce the amount of neuraxial pain medication required for comfort. For the study, Acetaminophen or placebo capsules will be administered at the time of neuraxial analgesia placement and then administered every 6 hours until delivery. Overall consumption of neuraxial pain medication will be determined.

DETAILED DESCRIPTION:
Acetaminophen 1000 mg or placebo capsules will be administered at the time of neuraxial analgesia placement and continued every 6 hours until delivery. Vital signs, scores for pain, nausea, itching, and sleepiness will be also obtained. Evaluation of consumption of neuraxial analgesic medication will be included in the final analysis for the differences between the 2 groups

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age not allergic to study medications

Exclusion Criteria:

* pre-eclampsia in labor AND with demonstrated significant abnormal liver enzyme function changes non-English speaking subjects

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Pan, MD, MSEE, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were approached after being admitted to the labor and delivery unit of our facility about participation in this clinical trial
Groups:
- Acetaminophen: 1000 mg every 6 hours during labor up to maximum 3 doses
  Acetaminophen: administered every 6 hours by mouth up to 3 doses
- Placebo: placebo capsule identical to the acetaminophen capsule will be administered every 6 hours to a maximum of 3 doses
  Placebo
Period: Overall Study
Arm/Group | Acetaminophen | Placebo
Started | 14 | 19
Completed | 12 | 15
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Placebo | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 7 | 11 | 18
  african american | 5 | 2 | 7
  hispanic | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Neuraxial Analgesic Drug Consumption Per Hour
Description: subject evaluated every 2 hours with the amount of neuraxial analgesia consumed during that time period. Study med administered up to 24 hours. labor analgesia continue until delivery.
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 12 | 15
milliliters | 155.19 (109.56) | 143.41 (73.48)
Statistical Analysis 1: Comparison: Acetaminophen; Test type: Other — unpaired t-test compared between groups; p > 0.05, unpaired t-test compared between groups
Statistical Analysis 2: Comparison: Placebo; Test type: Other — unpaired t-test compared between groups; p > 0.05, unpaired t-test compared between groups

ADVERSE EVENTS:
Time Frame: information collected up to 24 hours after the initiation of neuraxial analgesia
Arm/Group | Acetaminophen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes